CLINICAL TRIAL: NCT02335086
Title: DNA Damage and Repair Proteins In Patients With Atherosclerotic Coronary Artery Disease
Brief Title: DNA Damage & Repair Proteins In Patients With Atherosclerotic Coronary Artery Disease
Acronym: DECODE
Status: Completed | Type: Observational
Sponsor: University of Surrey (Other)
Collaborators: Ashford and St. Peter's NHS Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: 13/LO/0238
Record Dates: First submitted 2014-10-28; First posted 2015-01-09 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Coronary Atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, serum, white blood cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Stable angina patients: Patients with stable angina not responding to 2 anti-anginals presenting for coronary angiography with the possibility of proceeding to stent implantation at Ashford and St. Peter's Hospital.
  Clinical and angiographic exclusion criteria as stated in the study protocol.
- NSTEMI patients: Patients presenting to Ashford and St. Peter's Hospital with an non ST-elevation myocardial infarction defined by :
  Detection of a rise and/or fall of cardiac biomarker values (troponin I) with at least one value above the 99th percentile upper reference limit at analysing laboratories at Ashford and St. Peter's Hospital along with at least one of the following:
  * Symptoms of ischaemia
  * Development of pathologic Q waves in the electrocardiogram (ECG)
  * New or presumed new significant ST-segment-T wave (ST-T) changes on ECG.
  * Identification of an intracoronary thrombus by angiography.
  * Imaging evidence of new loss of viable myocardium or a new regional wall motion abnormality.

SUMMARY:
The purpose of this study is:

1. To examine the association between stable and unstable coronary artery disease (CAD) with markers of DNA damage and repair,
2. To examine the association between plaque morphology as assessed by frequency-domain optical coherence tomography (FD-OCT) and markers of DNA damage and repair in order to identify potential markers of plaque instability,
3. To examine the association between markers of DNA damage and repair and major adverse cardiovascular events defined as death, MI and unplanned percutaneous or surgical revascularization,

DETAILED DESCRIPTION:
Hypotheses ----------------

We hypothesise that defective DNA damage response is an important aetiological factor in the development of CAD, underlying CAD severity and development. If this hypothesis is true, then we predict that:

1. There is differential expression of markers of DNA damage and repair in patients with stable angina, a model of stable CAD, and patients with non ST-elevation myocardial infarction (NSTEMI), a model of unstable CAD.
2. Differential expression of markers of DNA damage and repair correlate with plaque morphology and stability as defined by FD-OCT,
3. Markers of DNA damage and repair can serve as distinguishing markers of stable and unstable CAD,

   Methodology

   ------------------

   Study Population:

   Patients presenting with stable angina undergoing percutaneous revascularization at Ashford and St. Peter's Hospitals Foundation Trust will be prospectively enrolled. Data regarding demographic, clinical, and procedural characteristics of patients will be collected by the Ashford and St. Peter's Hospitals Foundation Trust research personnel and entered into a secure, encrypted, dedicated database.

   Pre-defined clinical and angiographic inclusion and exclusion criteria will be met as per the DECODE study protocol.

   FD-OCT (St. Jude Medical ILUMIEN OCT System) will be performed in all the three main epicardial coronary arteries prior to target vessel PCI after administration of glyceryl trinitrate. Data will be acquired in a designated, secure compute and sent to a corelab for analysis. Quantitative measurements will include endoluminal area, plaque area, as well as plaque parameters including thin- capped fibroatheromas (TCFA), fibrous tissue, lipid core and calcium. TCFA will be defined by lipid-rich plaque with cap thickness ≤ 65μm.

   Culprit lesions will be defined according to electrocardiographic criteria (ST-segment shift or T-wave inversion) and angiographic appearances (luminal irregularities consistent with lesion ulceration, filling defect(s) consistent with thrombus, or point of angiographic maximal stenosis) in patients with NSTEMI and angiographic stenosis ≥ 70% in patients with stable angina not responding to at least two anti-anginal medications.

   Blood will be drawn immediately prior to percutaneous coronary intervention. In addition to routine haematological and biochemical parameters (complete blood count, white cell count, platelet count, creatinine, urea, sodium, potassium, cholesterol, glucose, troponine I, creatinine phosphokinase, liver function tests and clotting screen) one additional blood sample will be taken and separated into plasma and serum. Polymorphonuclear leukocytes will be used for measurements of DNA damage and repair proteins.

   Clinical follow-up will occur at 30-day and 12-month from enrolment by telephone interview and clinic visits. A repeat blood sample will be taken for analysis of DNA damage and repair proteins.

   DNA Damage

   ------------------

   DNA damage will be analysed by measuring DNA strand breaks in cell pellets using the comet assay. Serum oxidised purines will also be measured using an ELISA based assay. The transcriptional activation of DNA damage proteins will be assessed by real time PCR. For this, RNA will be isolated using a Roche High Pure Isolation kit. The RT2 First Strand Kit (SABioscience) will be utilised for reverse transcription of total RNA. Automated PCR will be set up and the raw data will be normalised using the average cycle threshold (ct) value of four housekeeping genes (B2M, RPL13A, GAPDH, and ACTB).

   Whether differential gene expression leads to differential protein expression will be determined by Western blotting. Moreover, the phosphorylation status of DNA damage proteins will also be assessed.

   DNA repair activity will also be assessed for several DNA repair enzymes important for the repair of base damage generated by reactive oxygen and nitrogen species. DNA repair activity will be measured by using in-vitro oligonucleotide-based cleavage assays.

   Finally, we will then correlate measures of DNA damage and repair with patient presentation (stable angina vs. NSTEMI), MACE, and FD-OCT derived parameters including the number of TCFA, plaque volume and percentage of plaque components.

   Statistical analysis

   -------------------------

   Statistical analysis will be performed using SAS version 8.2 (SAS institute Inc., Cary, North Carolina). Biomarker parameters will be tested for an association with patient presentation (stable angina vs. NSTEMI) and MACE using a log-rank test. OCT derived parameters will be tested for an association with biomarkers using univariate Cox proportional hazard regression. Parameters with a significance level of ≤0.1 on univariate analysis will undergo multivariate Cox proportional hazard analysis. A p value <0.05 will be considered statistically significant.

   The recruitment period is anticipated to last 15-18 months, with data collation and interpretation throughout recruitment and analysis anticipated to be complete by 24 months.

ELIGIBILITY:
Inclusion Criteria

-----------------------

Clinical:

1. Age ≥ 18 years
2. Stable angina not responding to at least two anti-anginal medications (beta blockers, calcium channel antagonists, long acting nitrate, Nicorandil, Ivabradine, or Ranolazine), or NSTEMI.
3. Patient is able to provide written, informed consent and is able to follow protocol procedures.

Angiographic:

1. Successful and uncomplicated percutaneous coronary intervention (PCI) performed in the major epicardial coronary arteries.

NB: Successful PCI is defined as residual diameter stenosis < 5% in all treated lesions with thrombolysis in myocardial infarction (TIMI)-3 flow (defined as normal flow which fills the distal coronary bed completely), absence of intraprocedural chest pain or ST-segment changes lasting > 10 minutes, persistent vessel closure, no re-flow, perforation, dissection or requirement for cardiopulmonary resuscitation, defibrillation, pacemaker or intra-aortic balloon implantation.

Exclusion Criteria:

------------------------

Clinical:

1. Presentation with ST-elevation MI (STEMI),
2. Decompensated heart failure, hypotension, shock, refractory ventricular tachycardia, acute conduction disorders, left ventricular ejection fraction ≤ 30%,
3. Prior coronary revascularization,
4. Any form of surgery up to three months prior to enrolment,
5. Active inflammatory disorders,
6. Bleeding diathesis,
7. Known allergy, hypersensitivity, or contraindication to aspirin, heparin, or thienopyridines,
8. Life expectancy less than 1 year,
9. Diabetes mellitus.

Angiographic:

1. Left main coronary artery stenosis ≥ 50%,
2. Coronary artery bypass surgery planned within one year of the PCI,
3. Anatomical conditions precluding three-vessel FD-OCT (significant tortuosity, severe calcification, chronic total occlusion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting with stable angina (n=50) or NSTEMI (n=50) undergoing percutaneous revascularization at Ashford and St. Peter's Hospitals Foundation Trust will be prospectively enrolled. Data regarding demographic, clinical, and procedural characteristics of patients will be collected by the Ashford and St. Peter's Hospitals Foundation Trust research personnel and entered into a secure, dedicated database. Results will be compared to age and sex matched controls
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2014-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Difference in DNA ligase activity in peripheral blood mononuclear cells of patients with stable angina and non-ST-elevation myocardial infarction | 18 months
  DNA ligase (DNA repair enzyme) activity measured using units per well, in peripheral mononuclear cells between stable and NSTEMI patients undergoing percutaneous coronary intervention.

SECONDARY OUTCOMES:
Plaque fibrous cap thickness and its association with major adverse cardiovascular events (MACE) | 18 months
  Examine the correlation between markers of DNA damage with plaque morphology and cap thickness, measured in micrometres, as assessed with optical coherence tomography and major adverse cardiac events defined as a composite of death, MI and target lesion revascularisation.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Ashford and St. Peter's Hospital, Chertsey, Surrey
  - University of Surrey, Guildford, Surrey

REFERENCES:
- [Derived] Dan K, Garcia-Garcia HM, Yacob O, Kuku KO, Kolm P, Shah N, Bennett MR, Curzen N, Waksman R, Mahmoudi M. Comparison of plaque distribution and wire-free functional assessment in patients with stable angina and non-ST elevation myocardial infarction: an optical coherence tomography and quantitative flow ratio study. Coron Artery Dis. 2021 Mar 1;32(2):131-137. doi: 10.1097/MCA.0000000000000944. PMID 32826449
- [Derived] Shah N, Meira LB, Elliott RM, Hoole SP, West NE, Brown AJ, Bennett MR, Garcia-Garcia HM, Kuku KO, Dan K, Kolm P, Mariathas M, Curzen N, Mahmoudi M. DNA Damage and Repair in Patients With Coronary Artery Disease: Correlation With Plaque Morphology Using Optical Coherence Tomography (DECODE Study). Cardiovasc Revasc Med. 2019 Sep;20(9):812-818. doi: 10.1016/j.carrev.2019.04.028. Epub 2019 May 23. PMID 31178349